CLINICAL TRIAL: NCT04789031
Title: Muscle Status to Oral Nutritional Supplementation in Hemodialysis Patients With Protein Energy Wasting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taylor's University (Other)
Collaborators: National Kidney Foundation, United States (Other)
Responsible Party: Principal Investigator, Tilakavati Karupaiah, Prof Dr Tilakavati Karupaiah, Taylor's University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NKF/2018/SBS/01; NMRR-16-2525-32068 (Registry Identifier: National Medical Research Register)
Record Dates: First submitted 2021-03-01; First posted 2021-03-09 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Muscle Wasting; End Stage Renal Disease on Dialysis
Keywords: hemodialysis; protein energy wasting; oral nutritional supplementation; ultrasound imaging
MeSH Terms: conditions — Muscular Atrophy | interventions — Dietary Supplements

STUDY DESIGN:
Intervention Model Description: Patients were allocated to intervention and control group. The intervention group received commercial renal-specific ONS for six months. Both groups received standard nutritional counseling during the study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients received oral nutritional supplementation and standard nutritional counseling for 6 months.
  Interventions: Dietary Supplement: Oral nutritional supplementation (ONS)
- Control group (No Intervention): Patients received standard nutritional counseling for 6 months.

INTERVENTIONS:
Dietary Supplement: Oral nutritional supplementation (ONS) — Patients received a renal specific ONS (Novasource Renal, Nestle) providing 475 kcal and 21.7g of protein per serving on a daily basis for 6 months. This was a ready-to- drink formula available in a tetrabrik pack. Patients consumed the product 30 minutes after commencing their dialysis session or at home after completion of dialysis.
  Arms: Intervention group

SUMMARY:
This multi-centred randomized, open label-controlled trial consists of hemodialysis (HD) patients identified with protein energy wasting (PEW) using the International Society of Renal Nutrition and Metabolism criteria. Intervention provided was oral nutritional supplementation (ONS) for 6 months and changes in muscle status in response toward the treatment was measured using ultrasound imaging method pre- and post-intervention.

DETAILED DESCRIPTION:
This study is a multi-centred randomized, open label-controlled trial where a total of 54 HD patients (29 intervention; 27 control) with PEW were recruited from government, private and non-governmental organization settings. Patients were randomized to either the intervention or control group. The intervention group received ONS (475 kcal and 21.7 g of protein), daily for 6 months. Both intervention and control group received standard nutritional counseling during the study period.

Patients who consented were subjected to a screening for identification of PEW and other eligibility criteria. Patients who fulfilled the inclusion criteria were randomized to either control or intervention group. During the 6 months of treatment period, patients in both control and intervention groups were assessed at baseline, 3rd months and 6th months for changes in muscle status using ultrasound imaging and bio-impedance spectroscopy method, malnutrition inflammation complex syndrome using Malnutrition-Inflammation Score, and other measures indicative of nutritional status including anthropometry, biochemistry, dietary intake and quality of life assessment. These parameters were compared at baseline and 6 months for within and between group differences using general linear model test.

ELIGIBILITY:
Inclusion Criteria:

* HD patients receiving standard dialysis treatment (3 sessions per week, 4 hours per session) for >3 months
* Aged between 18 to 70 years old
* Diagnosed with PEW using the ISRNM criteria

Exclusion Criteria:

* History of poor adherence to HD treatment
* Prolonged hospitalization or surgery in the past 3 months prior to recruitment
* Diagnosed with inflammatory diseases or malignancy
* Vegetarian
* Regular intake of ONS

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Changes in muscle status | Baseline versus 6 months
  Effect of ONS on improving muscle status using ultrasound imaging (quadriceps muscle thickness and cross-sectional area of the rectus femoris muscle) and bio-impedance spectroscopy method (measuring lean tissue mass)

SECONDARY OUTCOMES:
Changes in malnutrition-inflammation complex syndrome | Baseline versus 6 months
  Effect of ONS on improving malnutrition complex syndrome using Malnutrition-Inflammation Score (questionnaire) with lower ratings indicating well-nourished
Changes in anthropometric measures | Baseline versus 6 months
  Effect of ONS on improving post-dialysis weight and body mass index
Changes in nutrition-related biochemistry measures | Baseline versus 6 months
  Effect of ONS on improving serum albumin and serum prealbumin levels
Changes in dietary parameters | Baseline versus 6 months
  Effect of ONS on improving dietary energy and protein intake assessed using 24-hour diet recall forms
Changes in quality of life | Baseline versus 6 months
  Effect of ONS in improving quality of life assessed using the short form-36 questionnaire, with higher total score indicating better quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Tilakavati Karupaiah, PhD, Principal Investigator — Taylor's University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carrero JJ, Thomas F, Nagy K, Arogundade F, Avesani CM, Chan M, Chmielewski M, Cordeiro AC, Espinosa-Cuevas A, Fiaccadori E, Guebre-Egziabher F, Hand RK, Hung AM, Ikizler TA, Johansson LR, Kalantar-Zadeh K, Karupaiah T, Lindholm B, Marckmann P, Mafra D, Parekh RS, Park J, Russo S, Saxena A, Sezer S, Teta D, Ter Wee PM, Verseput C, Wang AYM, Xu H, Lu Y, Molnar MZ, Kovesdy CP. Global Prevalence of Protein-Energy Wasting in Kidney Disease: A Meta-analysis of Contemporary Observational Studies From the International Society of Renal Nutrition and Metabolism. J Ren Nutr. 2018 Nov;28(6):380-392. doi: 10.1053/j.jrn.2018.08.006. PMID 30348259
- [Background] Sahathevan S, Khor BH, Ng HM, Gafor AHA, Mat Daud ZA, Mafra D, Karupaiah T. Understanding Development of Malnutrition in Hemodialysis Patients: A Narrative Review. Nutrients. 2020 Oct 15;12(10):3147. doi: 10.3390/nu12103147. PMID 33076282
- [Background] Fouque D, Kalantar-Zadeh K, Kopple J, Cano N, Chauveau P, Cuppari L, Franch H, Guarnieri G, Ikizler TA, Kaysen G, Lindholm B, Massy Z, Mitch W, Pineda E, Stenvinkel P, Trevino-Becerra A, Wanner C. A proposed nomenclature and diagnostic criteria for protein-energy wasting in acute and chronic kidney disease. Kidney Int. 2008 Feb;73(4):391-8. doi: 10.1038/sj.ki.5002585. Epub 2007 Dec 19. PMID 18094682
- [Background] Ikizler TA, Cano NJ, Franch H, Fouque D, Himmelfarb J, Kalantar-Zadeh K, Kuhlmann MK, Stenvinkel P, TerWee P, Teta D, Wang AY, Wanner C; International Society of Renal Nutrition and Metabolism. Prevention and treatment of protein energy wasting in chronic kidney disease patients: a consensus statement by the International Society of Renal Nutrition and Metabolism. Kidney Int. 2013 Dec;84(6):1096-107. doi: 10.1038/ki.2013.147. Epub 2013 May 22. PMID 23698226
- [Background] Liu PJ, Ma F, Wang QY, He SL. The effects of oral nutritional supplements in patients with maintenance dialysis therapy: A systematic review and meta-analysis of randomized clinical trials. PLoS One. 2018 Sep 13;13(9):e0203706. doi: 10.1371/journal.pone.0203706. eCollection 2018. PMID 30212514
- [Background] Sahathevan S, Khor BH, Singh BKS, Sabatino A, Fiaccadori E, Daud ZAM, Ali MS, Narayanan SS, Tallman D, Chinna K, Goh BL, Gafor AHA, Ahmad G, Morad Z, Khosla P, Karupaiah T, On Behalf Of The Patch Study Malaysia Investigators. Association of Ultrasound-Derived Metrics of the Quadriceps Muscle with Protein Energy Wasting in Hemodialysis Patients: A Multicenter Cross-Sectional Study. Nutrients. 2020 Nov 23;12(11):3597. doi: 10.3390/nu12113597. PMID 33238633
- [Background] Sabatino A, Regolisti G, Delsante M, Di Motta T, Cantarelli C, Pioli S, Grassi G, Batini V, Gregorini M, Fiaccadori E. Noninvasive evaluation of muscle mass by ultrasonography of quadriceps femoris muscle in End-Stage Renal Disease patients on hemodialysis. Clin Nutr. 2019 Jun;38(3):1232-1239. doi: 10.1016/j.clnu.2018.05.004. Epub 2018 May 19. PMID 29866494
- [Background] Mah JY, Choy SW, Roberts MA, Desai AM, Corken M, Gwini SM, McMahon LP. Oral protein-based supplements versus placebo or no treatment for people with chronic kidney disease requiring dialysis. Cochrane Database Syst Rev. 2020 May 11;5(5):CD012616. doi: 10.1002/14651858.CD012616.pub2. PMID 32390133
- [Background] Lu Y, Wang YJ, Lu Q. The effect of oral nutritional supplement on muscle fitness of patients undergoing dialysis: A systematic review and meta-analysis. J Adv Nurs. 2021 Apr;77(4):1716-1730. doi: 10.1111/jan.14684. Epub 2020 Dec 3. PMID 33270269
- [Derived] Sahathevan S, Karupaiah T, Khor BH, Sadu Singh BK, Mat Daud ZA, Fiaccadori E, Sabatino A, Chinna K, Abdul Gafor AH, Bavanandan S, Visvanathan R, Yahya R, Wahab Z, Goh BL, Morad Z, Bee BC, Wong HS. Muscle Status Response to Oral Nutritional Supplementation in Hemodialysis Patients With Protein Energy Wasting: A Multi-Center Randomized, Open Label-Controlled Trial. Front Nutr. 2021 Dec 10;8:743324. doi: 10.3389/fnut.2021.743324. eCollection 2021. PMID 34977109